CLINICAL TRIAL: NCT01270724
Title: A Phase II Clinical Trial of Induction Chemotherapy Regimen Gemcitabine, Paclitaxel and Oxaliplatin (GemPOx) Followed by a Single Cycle of High Dose Chemotherapy (HDC) and Autologous Hematopoietic Stem Cell Rescue (AuHSCR) for Patients With Recurrent or Progressive Intracranial Germ Cell Tumors
Brief Title: Gemcitabine, Paclitaxel and Oxaliplatin (GemPOx)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GemPOx
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Results first posted 2025-10-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: CNS Germ Cell Tumor
MeSH Terms: interventions — Gemcitabine; Paclitaxel; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine, Paclitaxel and Oxaliplatin (GemPOx) (Experimental): Two to four cycles of induction therapy with open label GemPOx followed by consolidation and autologous stem cell transplant (ASCT).
  Interventions: Drug: Gemcitabine, Paclitaxel and Oxaliplatin (GemPOx).

INTERVENTIONS:
Drug: Gemcitabine, Paclitaxel and Oxaliplatin (GemPOx). — Two to four cycles of induction therapy with GemPOx followed by consolidation and ASCT.
  Other Names: GemPOx

SUMMARY:
This study will look to see how well patients with relapsed or recurrent intracranial germ cell tumors respond to the new combination of chemotherapy (in induction)of Gemcitabine, Paclitaxel and Oxaliplatin (GemPOx) followed by consolidation chemotherapy and autologous stem cell rescue.

ELIGIBILITY:
Inclusion Criteria:

* ICGCT including pure germinoma and MMGCT.
* Patients with histologically proven germinoma and MMGCT, including endodermal sinus tumor (yolk sac tumor), embryonal carcinoma, choriocarcinoma and mixed germ cell tumor will be eligible for the study.
* Patients with mature/immature teratoma who have tumor marker elevations are eligible on this study.
* Patient with ONLY mature and/or immature teratoma are ineligible in the absence of the tumor marker elevations.

Exclusion Criteria:

* Patients with ICGCTs who are newly diagnosed are excluded from the study.
* Patients with the diagnosis of mature or immature teratoma in the absence of tumor marker elevations are excluded from the study.
* Patients who are pregnant or breastfeeding are excluded from the study.
* Patients who have received previously a high dose chemotherapy regimen and autologous transplant are excluded from this study.
* Patients who have received gemcitabine, oxaliplatin and/or paclitaxel are excluded from this study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-08; Primary Completion 2019-10-23 (Actual); Study Completion 2019-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randal Olshefski, MD, Principal Investigator — Nationwide Children's Hospital
Locations (5):
- United States (5):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - New York University Langone Medical Center, New York, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - The Ohio State University Wexner Medical Center_The James Comprehensive Cancer Center, Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Nine patients with confirmed relapsed or refractory intracranial GCT were enrolled after signing informed consent, and received at least two cycles of GemPOx, of which all but one had relapsed or refractory NGGCTs. One patient with progressive disease was found to have pathologically confirmed malignant transformation to pure embryonal rhabdomyosarcoma (without GCT elements), hence was ineligible and not included in the analysis.
Period: Overall Study
Arm/Group | Gemcitabine, Paclitaxel and Oxaliplatin (GemPOx)
Started (2009) | 10 (12/21/2009 - Study IRB approved at CHLA.)
2012 | 6 (1 patient was later deemed ineligible bases on pathology and was taken off study.)
2013 | 1 (1 enrollment in 2013.)
2014 | 1 (1 enrollment in 2014.)
2016 | 1 (1 enrollment in 2016.)
2017 | 1 (1 enrollment in 2017.)
Completed | 7 (10/23/2019 - Study closed to accrual in NCH IRB.)
Not Completed | 3

BASELINE CHARACTERISTICS:
Groups:
- Gemcitabine, Paclitaxel and Oxaliplatin (GemPOx): Two to four cycles of induction therapy with open label GemPOx followed by consolidation and autologous stem cell transplant (ASCT).
  Gemcitabine, Paclitaxel and Oxaliplatin (GemPOx).: Two to four cycles of induction therapy with GemPOx followed by consolidation and ASCT.
  Nine patients with confirmed relapsed or refractory intracranial GCT were enrolled after signing informed consent, and received at least two cycles of GemPOx, of which all but one had relapsed or refractory NGGCTs. One patient with progressive disease was found to have pathologically confirmed malignant transformation to pure embryonal rhabdomyosarcoma (without GCT elements), hence was ineligible and not included in the analysis. Patients who experienced sufficient responses proceeded to receive HDCx with AuHPCR. Treatment response was determined based on radiographic tumor assessments and tumor markers.
Arm/Group | Gemcitabine, Paclitaxel and Oxaliplatin (GemPOx)
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants] — Population: 10 patients were consented and enrolled on therapy; one patient was declared ineligible on path review therefore not included in the final analysis or manuscript. 9 patients total will be included in final analyses.
  Participants
    <=18 years | 5
    Between 18 and 65 years | 5
    >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 9
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 10
Patients enrolled on study with eligible diagnosis of CNS GCT including pure germinoma and MMGCT [Count of Participants; unit: Participants] | 9

OUTCOME MEASURES:

1. Primary Outcome: Response Rate
Description: To estimate response rate after at least two and up to four courses of induction chemotherapy with GemPOx regimen in patients with recurrent intracranial MMGCT
Time Frame: 16-32 weeks depending on individual patient response (remaining disease burden) to chemotherapy
Measure: Count of Participants; unit: Participants
Groups:
- Gemcitabine, Paclitaxel and Oxaliplatin (GemPOx): Gemcitabine, Paclitaxel and Oxaliplatin (GemPOx): Two to four cycles of induction therapy with GemPOx followed by consolidation and ASCT.
Arm/Group | Gemcitabine, Paclitaxel and Oxaliplatin (GemPOx)
Number analyzed (Participants) | 9
Participants
  CR, Complete Response | 0
  PR, Partial Response | 0
  SD, Stable Disease | 4
  PD, Progressive Disease | 2
  PR1, Partial Response with Normal Markers | 3
  PR2, Partial Response with Abnormal (but not rising) Markers | 0

2. Primary Outcome: The Rate of Completion of Induction Chemotherapy and Progression to High-dose Chemotherapy (HDC) With Autologous Hematopoietic Progenitor Cell Rescue (AuHPCR)
Time Frame: Mean follow-up of 44 months
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine, Paclitaxel and Oxaliplatin (GemPOx)
Number analyzed (Participants) | 9
Participants | 7

3. Secondary Outcome: OS and PFS
Description: To assess the overall survival (OS) and event-free survival (EFS) of patients treated on the GemPOx induction regimen followed by the HDC and AuHPCR in patients with progressive or recurrent CNS GCT.
  We hypothesize that specific CSF miRNA will prove to be accurate markers for tumor presence and predictors of response to therapy, with normalization being associated with improved progression-free survival (PFS) in patients under treatment for recurrent central nervous system (CNS) germ cell tumors (GCT).
Time Frame: 2 years, 3 years and 5 years
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Arm/Group | Gemcitabine, Paclitaxel and Oxaliplatin (GemPOx)
Number analyzed (Participants) | 9
Percentage of patients
  2-year PFS | 66.7 [28.2 to 87.9]
  3-year PFS | 55.6 [20.4 to 80.5]
  5-year PFS | 44.4 [13.6 to 71.9]
  2-year OS | 66.7 [28.2 to 87.9]
  3-year OS | 66.7 [28.2 to 87.9]
  5-year OS | 55.6 [20.4 to 80.5]

4. Post Hoc Outcome: Last Patient Follow-up Outcome
Description: The outcome of each patient at the last point of follow-up
Time Frame: Months in follow-up (up to 86 months follow-up)
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine, Paclitaxel and Oxaliplatin (GemPOx)
Number analyzed (Participants) | 9
Participants
  PR, Partial Response | 0
  SD, Stable Disease | 0
  PD, Progressive Disease | 0
  NED, No Evidence of Disease | 4
  DOD, Dead of Disease | 4
  Unknown, Lost to Follow-up | 1

ADVERSE EVENTS:
Time Frame: Each participant was followed for up to 5 months for adverse events (up to 4 cycles of Induction chemotherapy followed by one cycle of Consolidation therapy), or 30 days after the last dose of study drug was received. All-Cause Mortality was assessed for an average of 44 months
Arm/Group | Gemcitabine, Paclitaxel and Oxaliplatin (GemPOx)
All-Cause Mortality (participants affected / at risk) | 4/10
Serious Adverse Events (participants affected / at risk) | 2/10
Other Adverse Events (participants affected / at risk) | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine, Paclitaxel and Oxaliplatin (GemPOx) (N=10)
Death (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Death (General disorders) | 1 (1) — Encephalopathy
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine, Paclitaxel and Oxaliplatin (GemPOx) (N=10)
Allergic reaction (Immune system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
ALT (Investigations) | 1 (13) — The CRC wrote "ALT" but the only CTCAE term is Alanine aminotransferase increased - therefore, this is likely the true terminology
Anorexia (Metabolism and nutrition disorders) | 1 (1)
AST (Investigations) | 1 (7) — The CRC wrote "AST" but the only CTCAE term for this is Aspartate aminotransferase increased
Confusion (Psychiatric disorders) | 1 (1)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
GGT (Investigations) | 1 (1) — The CRC wrote "GGT" but the CTCAE term is "GGT increased"
Hemoglobin (Investigations) | 1 (1) — The CRC wrote "hemoglobin" but the CTCAE is "hemoglobin increased"
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2)
Hypernatremia (Metabolism and nutrition disorders) | 1 (4)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (3)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Infections and infestations, other (Infections and infestations) | 1 (2) — One of the two AEs says "fungal sepsis"
Low WBC (Investigations) | 1 (11) — The CRC wrote "Low WBC" but the CTCAE term is "White blood count decreased"
Lymphocyte count decreased (Investigations) | 1 (3)
Mucositis (Gastrointestinal disorders) | 1 (4) — Unknown location for mucositis based on CRC term
Neutropenia (Blood and lymphatic system disorders) | 1 (16)
Neutrophil count decreased (Investigations) | 1 (1)
Pain (Musculoskeletal and connective tissue disorders) | 1 (3)
Pain, oral (Gastrointestinal disorders) | 1 (2)
Platelet count decrease (Investigations) | 1 (8)
Ptosis (Eye disorders) | 1 (1) — CRC wrote "ptosis" but CTCAE lists "eyelid functioning disorder"

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-05): https://cdn.clinicaltrials.gov/large-docs/24/NCT01270724/Prot_SAP_000.pdf